CLINICAL TRIAL: NCT04489667
Title: HIV + Service Delivery and Telemedicine Through Effective PROs (+STEP)
Brief Title: HIV + Service Delivery and Telemedicine Through Effective PROs
Acronym: HIV+STEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not considered a clinical trial
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Eaton, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-300005613; 1R01MH124633-01 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-07-28 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: HIV/AIDS; Mental Health Issue; Substance Use Disorders
Keywords: Telemedicine; Patient reported outcomes; Focused training
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- +STEP Implementation (Other): All patients will receive +STEP as new standard of care at their clinic. This intervention will include staff training, PROs as part of routine care to screen for substance use and mental health disorders, and telemedicine for health care delivery.
  Interventions: Other: +STEP Implementation

INTERVENTIONS:
Other: +STEP Implementation — All patients receiving care at five RWHAP-funded clinics will receive the intervention (+STEP), in which patient-reported outcomes (PROs) on mental health and substance use disorder (SUD) will be integrated into routine care, targeted training will be provided for frontline clinicians on best practices for mental health and SUD treatment, and telemedicine for mental health and SUD will be offered to patients in need of expanded access to services.

SUMMARY:
This study will examine the impact of using a multicomponent intervention (patient reported outcomes, training, and telemedicine) to assist with the management of Mental Health (MH) and Substance Use Disorders (SUD) among people living with HIV (PLWH) engaged in care at UAB HIV Clinic, University of Alabama Family Clinic (Birmingham, AL), Thrive Federally Qualified Health Services Center (Huntsville), Health Services Center (Anniston), and Medical Advocacy and Outreach (Montgomery). The study will employ a hybrid type 2 implementation design. Because this intervention will be employed as the new standard of care at participating sites, all PLWH receiving care at the sites will receive this intervention. Patient-reported outcomes (PROs) will be integrated into routine care to screen PLWH for substance use and mental health disorders during routine clinical encounters. Training will be delivered to frontline clinicians so that they receive targeted knowledge on best practices for treatment of MH and SUD along with clinic-specific protocols for response to PROs on MH and SUD including treatment and referrals. Telemedicine services for MH and SUD will be offered to patients in need of expanded access to services due to a lack of clinic-level resources or additional barriers to traditional clinic visits such transportation, stigma, or substance using behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and receiving HIV care at one of the five participating sites

Exclusion Criteria:

* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing PROs | Baseline through Year 1
  We will quantify the percentage of patients completing a PRO related to mental health or substance use
Percentage of patients completing PROs | Year 1 through Year 2
  We will quantify the percentage of patients completing a PRO related to mental health or substance use
Percentage of patients completing PROs | Year 2 through Year 3
  We will quantify the percentage of patients completing a PRO related to mental health or substance use
Percentage of patients completing PROs | Year 3 through Year 4
  We will quantify the percentage of patients completing a PRO related to mental health or substance use
Percentage of patients completing PROs | Year 4 through Year 5
  We will quantify the percentage of patients completing a PRO related to mental health or substance use
Percentage of staff participating in training | Baseline through Year 1
  We will use attendance logs to determine how many staff at each site complete training
Percentage of staff participating in training | Year 1 through Year 2
  We will use attendance logs to determine how many staff at each site complete training
Percentage of staff participating in training | Year 2 through Year 3
  We will use attendance logs to determine how many staff at each site complete training
Percentage of staff participating in training | Year 3 through Year 4
  We will use attendance logs to determine how many staff at each site complete training
Percentage of staff participating in training | Year 4 through Year 5
  We will use attendance logs to determine how many staff at each site complete training
Percentage of patients receiving a referral to a mental health or substance use service | Baseline through Year 1
  We will use EMR and scheduling data to determine the number of referrals generated
Percentage of patients receiving a referral to a mental health or substance use service | Year 1 through Year 2
  We will use EMR and scheduling data to determine the number of referrals generated
Percentage of patients receiving a referral to a mental health or substance use service | Year 2 through Year 3
  We will use EMR and scheduling data to determine the number of referrals generated
Percentage of patients receiving a referral to a mental health or substance use service | Year 3 through Year 4
  We will use EMR and scheduling data to determine the number of referrals generated
Percentage of patients receiving a referral to a mental health or substance use service | Year 4 through Year 5
  We will use EMR and scheduling data to determine the number of referrals generated
Percentage of patients receiving mental health or substance use service based on attendance | Baseline through Year 1
  We will use EMR and scheduling data to determine the number of visits attended
Percentage of patients receiving mental health or substance use service based on attendance | Year 1 through Year 2
  We will use EMR and scheduling data to determine the number of visits attended
Percentage of patients receiving mental health or substance use service based on attendance | Year 2 through Year 3
  We will use EMR and scheduling data to determine the number of visits attended
Percentage of patients receiving mental health or substance use service based on attendance | Year 3 through Year 4
  We will use EMR and scheduling data to determine the number of visits attended
Percentage of patients receiving mental health or substance use service based on attendance | Year 4 through Year 5
  We will use EMR and scheduling data to determine the number of visits attended

SECONDARY OUTCOMES:
Percentage engaged in HIV care | Baseline through Year 1
  We will determine the number of participants engage in HIV care
Percentage engaged in HIV care | Year 1 through Year 2
  We will determine the number of participants engage in HIV care
Percentage engaged in HIV care | Year 2 through Year 3
  We will determine the number of participants engage in HIV care
Percentage engaged in HIV care | Year 3 through Year 4
  We will determine the number of participants engage in HIV care
Percentage engaged in HIV care | Year 4 through Year 5
  We will determine the number of participants engage in HIV care
Percentage receiving antiretroviral therapy for HIV | Baseline through Year 1
  We will determine the number of participants receiving HIV treatment
Percentage receiving antiretroviral therapy for HIV | Year 1 through Year 2
  We will determine the number of participants receiving HIV treatment
Percentage receiving antiretroviral therapy for HIV | Year 2 through Year 3
  We will determine the number of participants receiving HIV treatment
Percentage receiving antiretroviral therapy for HIV | Year 3 through Year 4
  We will determine the number of participants receiving HIV treatment
Percentage receiving antiretroviral therapy for HIV | Year 4 through Year 5
  We will determine the number of participants receiving HIV treatment
Number of Patients Achieving a Viral Load Suppression | Baseline through Year 1
  We will determine the number of participants who have achieved Viral Load suppression, s defined by a Viral load of <20 copies per milliliter
Number of Patients Achieving a Viral Load Suppression | Year 1 through Year 2
  We will determine the number of participants who have achieved Viral Load suppression, s defined by a Viral load of <20 copies per milliliter
Number of Patients Achieving a Viral Load Suppression | Year 2 through Year 3
  We will determine the number of participants who have achieved Viral Load suppression, s defined by a Viral load of <20 copies per milliliter
Number of Patients Achieving a Viral Load Suppression | Year 3 through Year 4
  We will determine the number of participants who have achieved Viral Load suppression, s defined by a Viral load of <20 copies per milliliter
Number of Patients Achieving a Viral Load Suppression | Year 4 through Year 5
  We will determine the number of participants who have achieved Viral Load suppression, s defined by a Viral load of <20 copies per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Eaton, MD, MSPH, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (5):
- United States (5):
  - Health Services Center, Anniston, Alabama
  - University of Alabama Family Clinic, Birmingham, Alabama
  - Thrive Federally Qualified Health Services Center, Huntsville, Alabama
  - Medical Advocacy and Outreach (MAO), Montgomery, Alabama
  - Unity Wellness Center, Opelika, Alabama

IPD SHARING:
Plan to Share IPD: Yes
The proposed project will comply with the NIH Data Sharing Policy, thus all data collected will be made available to outside investigators. To maintain HIPAA compliance, we will provide a limited-use dataset (i.e., stripped of identifying information). When possible, collaborative use of the data will be encouraged in order to enhance the quality of secondary analyses. Data will be made available as either a SPSS or Excel dataset, or as a tab-delimited ASCII file. Methods will be described through published papers, and relevant software and/or procedures documents.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data collected for this protocol will be made available to outside investigators in a timely fashion (defined by the NIH as no later than the acceptance of the primary outcome paper for publication)
Access Criteria: Requests for data will be handled on a case-by-case basis in consultation with the Co-Investigators and members of the team.

REFERENCES:
- [Background] Kozak MS, Mugavero MJ, Ye J, Aban I, Lawrence ST, Nevin CR, Raper JL, McCullumsmith C, Schumacher JE, Crane HM, Kitahata MM, Saag MS, Willig JH. Patient reported outcomes in routine care: advancing data capture for HIV cohort research. Clin Infect Dis. 2012 Jan 1;54(1):141-7. doi: 10.1093/cid/cir727. Epub 2011 Oct 31. PMID 22042879
- [Background] Mehrotra A, Huskamp HA, Souza J, Uscher-Pines L, Rose S, Landon BE, Jena AB, Busch AB. Rapid Growth In Mental Health Telemedicine Use Among Rural Medicare Beneficiaries, Wide Variation Across States. Health Aff (Millwood). 2017 May 1;36(5):909-917. doi: 10.1377/hlthaff.2016.1461. PMID 28461359
- [Background] Ickovics JR, Hamburger ME, Vlahov D, Schoenbaum EE, Schuman P, Boland RJ, Moore J; HIV Epidemiology Research Study Group. Mortality, CD4 cell count decline, and depressive symptoms among HIV-seropositive women: longitudinal analysis from the HIV Epidemiology Research Study. JAMA. 2001 Mar 21;285(11):1466-74. doi: 10.1001/jama.285.11.1466. PMID 11255423
- [Background] Springer SA, Dushaj A, Azar MM. The impact of DSM-IV mental disorders on adherence to combination antiretroviral therapy among adult persons living with HIV/AIDS: a systematic review. AIDS Behav. 2012 Nov;16(8):2119-43. doi: 10.1007/s10461-012-0212-3. PMID 22644066
- [Background] Sohail M, Rastegar J, Long D, Rana A, Levitan EB, Reed-Pickens H, Batey DS, Ross-Davis K, Gaddis K, Tarrant A, Parmar J, Raper JL, Mugavero MJ. Data for Care (D4C) Alabama: Clinic-Wide Risk Stratification With Enhanced Personal Contacts for Retention in HIV Care via the Alabama Quality Management Group. J Acquir Immune Defic Syndr. 2019 Dec;82 Suppl 3:S192-S198. doi: 10.1097/QAI.0000000000002205. PMID 31764254
- [Background] Powell BJ, McMillen JC, Proctor EK, Carpenter CR, Griffey RT, Bunger AC, Glass JE, York JL. A compilation of strategies for implementing clinical innovations in health and mental health. Med Care Res Rev. 2012 Apr;69(2):123-57. doi: 10.1177/1077558711430690. Epub 2011 Dec 26. PMID 22203646